CLINICAL TRIAL: NCT03251170
Title: Ketamine-based Versus Opioid-based for Rapid-sequence Induction of Anesthesia in Patients With Septic Shock
Brief Title: Ketamine Versus Fentanyl for Induction of Anesthesia in Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-12-2018
Record Dates: First submitted 2017-08-12; First posted 2017-08-16 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Ketamine; Fentanyl; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Experimental): This group of patients will receive: 1 mg/Kg ketamine + 0.05 mg/Kg midazolam for induction of anesthesia. Endotracheal tube will be inserted aided by 1 mg/Kg succinyl choline. Patients will undergo surgical procedure to eliminate the source of sepsis e.g. abdominal exploration. Invasive blood pressure monitor will be connected to the patient through an arterial catheter. Electrical velocimetry (cardiometry) device will be connected to the patient to measure cardiac output, stroke volume, and systemic vascular resistance.
  Interventions: Drug: Ketamine; Drug: Midazolam
- Fentanyl (Active Comparator): 2.5 mg/Kg fentanyl + 0.05 mg/Kg midazolam for induction of anesthesia. Endotracheal tube will be inserted aided by 1 mg/Kg succinyl choline. Patients will undergo surgical procedure to eliminate the source of sepsis e.g. abdominal exploration. Invasive blood pressure monitor will be connected to the patient through an arterial catheter. Electrical velocimetry (cardiometry) device will be connected to the patient to measure cardiac output, stroke volume, and systemic vascular resistance.
  Interventions: Drug: Fentanyl; Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Patients will receive :1 mg/Kg ketamine for induction of anesthesia
  Other Names: Katalar
  Arms: Ketamine group
Drug: Fentanyl — Patients will receive :2.5 mcg/Kg fentanyl for induction of anesthesia
  Arms: Fentanyl
Drug: Midazolam — Patients will receive 0.05 mg/Kg midazolam
  Other Names: Dormicum

SUMMARY:
The aim of this work is to compare two protocols (ketamine-midazolam versus fentanyl-midazolam) for induction of anesthesia in patients with septic shock aiming to find the most safe protocol with regards to hemodynamic status of patients

DETAILED DESCRIPTION:
Induction of anesthesia in hemodynamically compromised patients is a challenge for every anesthetist. Most of the intravenous induction agents have a negative effect on arterial blood pressure and cardiac output. Theoretically, the "ideal" emergency induction intravenous anesthetic should achieve rapid hypnosis and maintain the hemodynamic stability.

Ketamine has been reported as an induction anesthetic with a sympathomimetic activity. In patients with intact autonomic nervous system ketamine increases heart rate, cardiac output, and arterial blood pressure (ABP). Despite its sympathomimetic activity in hemodynamically stable patients, the hemodynamic response to ketamine in unstable cardiovascular conditions is not clear. No studies to the best of our knowledge compared Ketamine-based and opioid-based protocols in rapid sequence induction of anesthesia in hemodynamically unstable patients.

In this study, patients with severe sepsis or septic shock scheduled for surgery will be assigned to receive either ketamine or fentanyl for induction of anesthesia. After induction of anesthesia, endotracheal tube will be inserted aided by succinyl choline. Invasive blood pressure will be monitored through a transducer connected to arterial catheter. Electrical velocimetry (cardiometry) device will be used for non-invasive monitoring of cardiac output and stroke volume.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis patients
* With shock index (heart rate divided by systolic blood pressure) >0.7. or Sepsis patients with norepinephrine infusion.

Exclusion Criteria:

* Traumatic brain injury
* Cerebrovascular disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | 30 minutes after induction of anesthesia
  Mean arterial blood pressure measured by invasive transducer attached to arterial catheter

SECONDARY OUTCOMES:
cardiac output | 30 minutes after induction of anesthesia
  cardiac output measured in litres per minute measured by electrical velocimetry
Stroke volume | 30 minutes after induction of anesthesia
  cardiac stroke volume in milliliters measured by electrical velocimetry
heart rate | 30 minutes after induction of anesthesia
  heart rate measured in beat per minute
serum lactate | 30 minutes after induction of anesthesia
  serum lactate measured in mmol/liter
total norepinephrine dose | 30 minutes after induction of anesthesia
  total dose of norepinephrine measured in micrograms
Intra-operative inhalational anesthetic concentration | 30 minutes
  the concentration of inhalational anesthetic (%)
Incidence of post-induction hypotension | 5 minutes
  The percent of patients with severe hypotension after induction of anesthesia requiring stoppage of inhalational anesthesia or increasing the dose of vasopressors

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No